CLINICAL TRIAL: NCT03972527
Title: Photobiomodulation Therapy Using the MuReva Phototherapy System to Demonstrate Safety and Reduce the Incidence of Oral Mucositis in Adult Patients With Head and Neck Cancer Receiving Radiation Therapy With or Without Concurrent Chemotherapy
Brief Title: Photobiomodulation to Demonstrate Safety and Reduce the Incidence of Oral Mucositis in Adult Head & Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MuReva Phototherapy Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LLD-001
Record Dates: First submitted 2019-05-28; First posted 2019-06-03 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Oral Mucositis (Ulcerative); Oral Mucositis (Ulcerative) Due to Radiation; Oral Mucositis (Ulcerative) Due to Antineoplastic Therapy; Head and Neck Cancer
Keywords: photobiomodulation; LLLT (low-level laser therapy); low-level laser therapy; oral mucositis; wound healing; radiation therapy; chemotherapy; antineoplastic therapy; side effects; phototherapy; low-level light therapy
MeSH Terms: conditions — Stomatitis; Ulcer; Head and Neck Neoplasms | interventions — Low-Level Light Therapy; Analgesia; Acetaminophen; Mouthwashes

STUDY DESIGN:
Intervention Model Description: A prospective, multi-center, randomized, double-blind, placebo controlled, adaptive sample size, two-treatment parallel, pivotal clinical study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The sponsor, clinical research organization (CRO), subjects, research staff and Investigators performing the weekly OM evaluations for the study will be blinded to the treatment assignments. Subjects will be mandated to use light-blocking eyewear.
  Only the research staff delivering treatment will be unblinded. No other personnel or visitors will be allowed in the treatment room during active/sham treatment.
  The Investigators will not administer the daily treatment and will not visit or observe the patient during device use in order to remain blinded. The Investigators will also remain blinded to the patients' responses to the weekly Self-Assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Active Device Treatment Cohort - Chemoradiation therapy (Active Comparator): The MuReva Phototherapy System consists of Light Control Unit and two Mouthpiece Cable Assemblies. Subjects will begin device treatment photobiomodulation sessions on the first day of radiotherapy (RT) treatment. They will receive once-daily investigative device photobiomodulation treatments prior to radiation therapy (RT) with their assigned Mouthpiece for 5 days per week for the duration of their CRT treatment. Each device treatment session will last up to 5 minutes, not including up to 5 additional minutes for treatment breaks. All subjects will visit the study site once during the Screening period (Days -28 to 1) and an anticipated 30 to 40 times during the treatment period. Each patient will be assigned their own Mouthpiece Cable Assembly set.
  Interventions: Device: Photobiomodulation; Other: Routine Oral Care and Analgesia
- Sham Device Treatment Cohort- Chemoradiation therapy (Sham Comparator): The MuReva Phototherapy System (or sham control) is a Light Control Unit and a set of Mouthpiece Cable Assemblies. The sham control Mouthpiece Cable Assemblies will appear identical to the active Mouthpiece Cable Assembly, and will be used in the same manner as the active cohort. However, the sham control device will be configured where the mouthpiece will not emit any light at any time during the study. The same Light Control Unit will be used with sham and active Mouthpiece Cable Assemblies. Each patient will be assigned their own Mouthpiece Cable Assembly set.
  Interventions: Other: Routine Oral Care and Analgesia
- Active Device Treatment Cohort - Radiation therapy only (Active Comparator): The MuReva Phototherapy System consists of Light Control Unit and two Mouthpiece Cable Assemblies. Subjects will begin device treatment photobiomodulation sessions on the first day of radiotherapy (RT) treatment. They will receive once-daily investigative device photobiomodulation treatments prior to radiation therapy (RT) with their assigned Mouthpiece for 5 days per week for the duration of their CRT treatment. Each device treatment session will last up to 5 minutes, not including up to 5 additional minutes for treatment breaks. All subjects will visit the study site once during the Screening period (Days -28 to 1) and an anticipated 30 to 40 times during the treatment period. Each patient will be assigned their own Mouthpiece Cable Assembly set.
  Interventions: Device: Photobiomodulation; Other: Routine Oral Care and Analgesia
- Sham Device Treatment Cohort- Radiation therapy only (Sham Comparator): The MuReva Phototherapy System (or sham control) is a Light Control Unit and a set of Mouthpiece Cable Assemblies. The sham control Mouthpiece Cable Assemblies will appear identical to the active Mouthpiece Cable Assembly, and will be used in the same manner as the active cohort. However, the sham control device will be configured where the mouthpiece will not emit any light at any time during the study. The same Light Control Unit will be used with sham and active Mouthpiece Cable Assemblies. Each patient will be assigned their own Mouthpiece Cable Assembly set.
  Interventions: Other: Routine Oral Care and Analgesia

INTERVENTIONS:
Device: Photobiomodulation — Provide photobiomodulation therapy to subjects prior to each radiation therapy session.
  Other Names: low-level laser therapy
  Arms: Active Device Treatment Cohort - Chemoradiation therapy; Active Device Treatment Cohort - Radiation therapy only
Other: Routine Oral Care and Analgesia — Standard oral care, oral hygiene and oral pain protocols
  Other Names: Pain medication, oral rinses

SUMMARY:
The overall purpose of this clinical study is to evaluate safety and efficacy of the MuReva Phototherapy System with a light delivery mouthpiece to reduce the severity of oral mucositis (OM) in adult patients with squamous cell carcinoma of the oral cavity, oropharynx, tonsils and base of tongue receiving radiation therapy with or without concurrent chemotherapy.

DETAILED DESCRIPTION:
Study Design: A prospective, multi-center, randomized, double-blind, placebo controlled, adaptive sample size, two-treatment parallel, pivotal clinical study.

Protocol-eligible subjects will be randomized in a 1:1 allocation to receive either the active MuReva Phototherapy System or a sham control. Both the subjects and clinician evaluating the patients will be blinded to the treatment assignments. The sham device will be placed in the patient's mouth and operated in the same manner as the active device, but not deliver any therapy.

Subjects will begin device treatment sessions on the first day of radiation treatment (RT) and will continue to receive once daily treatments prior to RT with their assigned device for 5 days per week for the duration of their RT treatment (approximately 6 to 8 weeks, for a total of 30 to 40 device sessions depending on the standard of care regimen for the type of cancer). Each device treatment session will last approximately 10 minutes in total. Light therapy parameters for the MuReva Phototherapy System will be as follows for all subjects receiving active light therapy: 660nm, 2-12 J/cm2 nominal fluence. Subjects who stay on RT treatment past 6 weeks will continue to receive treatment with their assigned devices up through 8 total weeks of treatment (for a maximum total of 40 phototherapy sessions). In addition, all subjects, regardless of randomization, will be kept on standard oral care, oral hygiene and oral pain protocols.

All subjects will visit the study site once during the Screening period (Days -28 to 1) and an anticipated 30 to 40 times during the treatment period (i.e., 5 days during each of the 6-8 RT treatment weeks). Weekly, subjects will be evaluated for oral mucositis and for device safety. The weekly assessments will continue through the final RT session. A post-therapy assessment will be done approximately 2 weeks after completion of RT. At the conclusion of this assessment each subject's participation in the study will be complete.

ELIGIBILITY:
INCLUSION CRITERIA

1. Subject has been diagnosed with pathologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, tonsil or base of tongue.
2. Within 28 days of Screening, subject is scheduled to receive a continuous course of Intensity-Modulated Radiation Therapy (IMRT) over an estimated 6 to 8 weeks (treatment week is defined as 5 fractions per week). The initial target volume encompassing the gross and subclinical disease sites will receive 5 fractions per week with a minimum cumulative dose of 50 Gray (Gy) for low to intermediate risk (sites of suspected subclinical spread) and maximum cumulative dose of 70 Gy for gross tumor volume/High risk (Primary tumor and involved lymph nodes).
3. The subject's planned radiation treatment fields include a minimum of 50 Gy to at least two oral cavity sites (i.e. buccal mucosa, floor of mouth, ventral tongue, lateral tongue, dorsal tongue, hard palate, and soft palate).
4. If the subject is receiving concurrent chemotherapy, the treatment plan includes Cisplatin administered in either a standard weekly (30-40 mg/m2) or approximately every 21 days (80-100mg/m2) regimen OR Carboplatin administered in standard weekly (1.0-2.0 AUC) regimen WITH/WITHOUT Paclitaxel administered in a standard weekly (30-45mg/m2) regimen.
5. Subject is at least 22 years of age.
6. Subject has no dental or oral health conditions that would preclude daily use of a mouthpiece and demonstrates capability in sustaining mouthpiece in oral cavity for recommended time during Screening procedure.
7. Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
8. Subject is able to read and understand the Informed Consent Form (ICF) and has voluntarily provided written informed consent.
9. For the entire duration of their treatment, the subject will not use any tobacco or nicotine products with the exception of nicotine patches.
10. For the entire duration of their treatment, the subject will not use any inhaled cannabis products or any illicit drugs.

EXCLUSION CRITERIA

1. Subject is currently receiving or has previously received chemotherapy or chemoradiotherapy within the past 2 years and the oral cavity has not yet fully recovered.
2. Subject is given neo-adjuvant or induction chemotherapy for Head and Neck cancer prior to starting RT.
3. Subject has been diagnosed with another type/site of cancer that has not been controlled.
4. Subject is pregnant or nursing.
5. Subject is receiving medications indicated for the treatment and/or prevention of mucositis (e.g., palifermin).
6. Subject has had prior radiation to the head and neck.
7. Subject has a diagnosis that is prone to affect wound healing, e.g., uncontrolled diabetes.
8. Subject has trismus with an interincisal distance of 30mm or less.
9. Subject has an active infection in the oropharynx and/or oral cavity (any infection in the oropharynx and/or oral cavity at the time of screening must be addressed prior to first radiation treatment).
10. Subject has a salivary disturbance, e.g., Sjögren's syndrome.
11. Subject has any grade of oral mucositis per WHO Oral Toxicity Scale.
12. Subject is receiving, or has received in the last 30 days, an investigational treatment, therapy, or medical device outside of this clinical study protocol.
13. Subject has a Baseline mouth pain score of greater than 5 out of 10 on question 6 of the OMWQ-HN. Exception can be made if Principal Investigator determines the cause of mouth pain is due to tumor or surgery site pain.
14. Subject is unable to participate in the study because of a concurrent or recent disease state that, in the opinion of the Principal Investigator, would affect the study endpoints, e.g., dental disease or COVID-19 (active or recovered).
15. Subject has 8 or more dental prostheses or implants.
16. Subject is not considered eligible at the discretion of the oral maxillofacial dentist/surgeon. Exception can be made if all items identified on the dental exam have been addressed prior to first radiation treatment.
17. Subject is receiving any medications with oral photoprotection indications.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
IThe primary effectiveness endpoint is the severity of oral mucositis at week 6 of radiation treatment according to the Oral Mucositis Index (OMI) score. | approximately 6 weeks after patient begins radiation therapy
  The primary effectiveness endpoint of the study is the severity of oral mucositis as assessed by the Oral Mucositis Index (OMI) score, on a scale of 0-60.

SECONDARY OUTCOMES:
World Health Organization (WHO) Oral Toxicity Scale at week 6 | approximately 6 weeks after patient begins radiation therapy
  The proportion of patients who have severe oral mucositis (Grade 3 or 4) at week 6 of treatment according to the World Health Organization (WHO) Oral Toxicity Scale.
Changes in overall quality of life over the 6-week treatment period | difference between baseline and (approximately) 6 weeks after patient begins radiation therapy
  Oral Mucositis Weekly Questionnaire-Head and Neck Cancer

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Oncology Institute, Long Beach, California
  - Miami Cancer Institute, Miami, Florida
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Erie County Medical Center, Buffalo, New York
  - NYU Langone, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - MetroHealth, Cleveland, Ohio
  - James Cancer Hospital at The Ohio State University, Columbus, Ohio
  - Oklahoma Cancer Specialtists and Research Intstitute, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify individual subjects. At most, the Web site will include a summary of the results after the study is completed. You can search this Web site at any time.
  If the results of this study are published, individual subject identity will remain confidential.
  Data, salivary fluid specimens and photographs collected in this research might be de-identified (name and any identifying information will be removed) and used for future research or distributed to another investigator for future research.
Supporting Information: SAP, CSR
Time Frame: December 2024 anticipated
Access Criteria: not yet determined